CLINICAL TRIAL: NCT06075901
Title: Reliability, Reproducibility and Performance Analysis of the Use of Tissue Flossing for Blood Flow Restriction.
Brief Title: Reliability and Performance Analysis of the Use of Tissue Flossing for Blood Flow Restriction.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, Principal investigator, Paulista University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FCT - UNESP
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hypertrophy; Muscle Strength
Keywords: tissue flossing; blood flow restriction
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood Flow Restriction with Cuffing (Active Comparator): The participant will use the Cuffing for Blood Flow Restriction training
  Interventions: Device: Blood Flow Restriction Cuff; Other: Training Protocol
- Blood Flow Restriction with Tissue Flossing (Experimental): The participant will use Tissue Flossing for Blood Flow Restriction training
  Interventions: Device: Tissue Flossing; Other: Training Protocol

INTERVENTIONS:
Device: Tissue Flossing — Tissue Flossing ia a elastic band that when applied exerts an external pressure above or below a muscle or joint of the extremities.
  Arms: Blood Flow Restriction with Tissue Flossing
Device: Blood Flow Restriction Cuff — Inflatable device that exerts an external pressure above a muscle or joint of the extremities.
  Arms: Blood Flow Restriction with Cuffing
Other: Training Protocol — The lower limb resistance training protocol will follow that recommended in the study by Patterson et al. for resistance training, and will last 4 weeks, with 3 training sessions per week, with a day break between sessions.

SUMMARY:
Blood flow restriction (RFS) is a widely studied technique that combines low-intensity exercise with vascular occlusion, resulting in muscular benefits. However, its application is challenging due to methodological variations and equipment costs. Tissue Flossing (TF) appears as an affordable alternative, but lacks solid scientific evidence.

DETAILED DESCRIPTION:
Objectives: to evaluate the intra- and inter-rater reliability of the occlusion pressure generated by TF, investigate the reproducibility of TF application on different days and compare TF with traditional RFS in terms of muscle gains.

Methods: the study is divided into two stages: First stage, randomized controlled crossover clinical trial, 80 healthy individuals aged 18 to 30 years old evaluated to determine the reliability of the TF. Participants will follow one of two types of randomization, with exclusions based on health criteria. Assessments include anthropometric characteristics, determination of occlusion pressure (POT), identification of 40% and 80% of POT, flow data and arterial diameter after TF application. Statistical analysis will use the intraclass correlation index (ICC) and specific models for intra- and inter-rater analyses. Second stage, randomized controlled clinical trial with parallel groups, 110 recreational athletes will be evaluated over four weeks. The initial procedures involve anthropometric assessments, POT determination, myotonometry, ultrasound, perceptual scale and 1RM test, applied to both lower limbs. Participants will perform a lower limb training protocol, using RFS and TF on different legs, following myotonometric and perceptual assessments. After training, final assessments will measure the same parameters initially assessed. Statistical analysis will use normality tests, Generalized Mixed Models and effect size analysis in SPSS software, with a significance level of p<0.05. Expected results: This study is expected to provide information on the reliability and reproducibility of TF in generating occlusion pressure. Furthermore, we seek to validate TF by comparing it with traditional RFS in terms of muscle gains. If effective, TF could become an affordable option to promote muscle gains, in different application scenarios.

Participants will be duly informed about the procedures and objectives of this study, and after agreeing, they will sign an informed consent form, effectively becoming part of it. In the consent form, participants will be asked if they agree to the use of their data if they choose to withdraw from the study. Participants will also be asked for permission for the research team to share relevant data with people at universities participating in the research or regulatory authorities, where relevant. The study will be sent for consideration and approval to the Research Ethics Committee of FCT/UNESP, Presidente Prudente, SP, Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who present one or more of the following characteristics will not be included:
* 1 presence of any health condition that contraindicates or prevents exercise;
* 2 diabetes and diagnosed high blood pressure;
* 3 inflammatory, psychiatric, cardiovascular and/or respiratory rheumatological disease; - -4 being dependent on alcohol, consuming drugs and/or being a smoker;
* 5 history of knee surgery (e.g., meniscal repair and ligament reconstruction) or recent lower limb musculoskeletal injury that may impair performance during tests or interventions (e.g., muscle injury, tendinopathy, patellofemoral pain and/or back pain column in the last six months);
* 6 use of ergogenic supplements to improve physical performance and/or muscle mass and/or vasoactive medications;
* 7 having one or more risk factors predisposing to thromboembolism

Exclusion Criteria:

* Participants will be excluded from the study if they:
* 1 have a health problem that does not allow them to continue;
* 2 wish to leave the study;
* 3 not sign the consent form

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Occlusion pressures (AOP, 80% and 40% of AOP) | First and Secund Stage - [Time Frame: baseline]
  To determine the AOP, the Doppler equipment transducer will be used, which will be positioned over the posterior tibial artery to capture the auscultatory pulse. A blood pressure cuff will be fixed to the participant's thigh close to the region of the inguinal fold of the dominant limb, and then with the inflatable region of the cuff on the medial portion of the thigh covering the femoral artery, it will be progressively inflated, waiting 15 seconds every 30 mmHg until the point at which the auscultatory pulse of the tibial artery is interrupted.
Assessment of arterial flow and diameter | First Stage - [Time Frame: baseline and all subsequent assessments]
  A Sonoline Sienna® vascular ultrasound will be used combined with a 40mm B-mode ultrasonic transducer with a 7.5 MHz linear beam, which will be coated with gel for acoustic contact and positioned longitudinally to the posterior tibial artery, enabling variables to be assessed. Doppler flow measurements of MI (peak systolic velocity [cm/s], end-diastolic velocity [cm/s] and arterial diameter).
Perceptual parameter | First and Secund Stage - [Time Frame: baseline and all subsequent assessments]
  The perceptual parameter will be evaluated using a Borg CR10+ scale, representing the perception of discomfort, 0 represents no discomfort and 10 extremely uncomfortable.
Tissue Flossing Assessment | First Stage - [Time Frame: The subsequent assessments]
  The application of tissue flossing on the leg will be carried out by always passing the elastic tape with 50% of the tape over the next strip, until the end of the elastic tape.
Weight | First and Secund Stage- [Time Frame: Baseline ]
  It will be collected with a weight balance
Height | First and Secund Stage- [Time Frame: Baseline ]
  It will be collected with a stadiometer
Body Fat | First and Secund Stage- [Time Frame: Baseline ]
  It will be collected with a adipometer
Arterial pressure | First and Secund Stage- [Time Frame: Baseline ]
  It will be collected with a sphygmomanometer
Perimetry of the dominant lower limb | First and Secund Stage- [Time Frame: Baseline ]
  It will be defined by the Waterloo Footedness
Limb length | First and Secund Stage- [Time Frame: Baseline ]
  Identified with a measuring tape
Perceived exertion scale | Secund Stage- [Time Frame: at the end of the training sessions]
  Adapted BORG scale, with 0 being "no effort" and 10 "maximum effort".
Method preference | Secund Stage- [Time Frame: final evaluation]
  Participants must answer a brief questionnaire about their preference for one of the RFS methods carried out, and justify why they chose it.
1 Maximum Repetition Test | Secund Stage- [Time Frame: baseline and final evaluation]
  The participant must be positioned seated on the extension chair with knees and feet hip-width apart, knees at 90° flexion determined by goniometry, hands holding the handles adjacent to the hips and lumbosacral spine in a firm position in contact with the back of the chair.
  1 repetition should be performed to familiarize the movement and 10 repetitions to warm up. At the beginning of the test, they will be instructed to maintain a movement pattern and avoid compensation. The RM is then defined by the highest load at which the participant is capable of performing 1 repetition without compensation.
Myotonometry | Secund Stage- [Time Frame: baseline during follow-up and final evaluation]
  Myotonometry will be assessed using the MyotonPRO® tool, which consists of a portable, wireless and non-invasive device.
  The measurement will be carried out once, and in each shot, the following myotonometry parameters will be calculated: the state of tension (tone) and biomechanical properties (rigidity and elasticity).
Ultrasound | Secund Stage- [Time Frame: baseline and final evaluation]
  The assessment of the muscular structure will be carried out using ultrasound images of the participant's lower limbs, which will be captured using BodyMetrix BX-2000.
  Participants will be assessed in the supine position with legs fully extended and muscles relaxed. The ultrasound transducer will be covered with water-soluble transmission gel and positioned perpendicular to the skin over the muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No